CLINICAL TRIAL: NCT07152964
Title: Clinical Correlation Between Medial Rectus Tendon Width and Surgical Dose Response in Commitant Esotropic Patients Undergoing Medical Rectus Recession
Brief Title: Medial Rectus Tendon Width and Surgical Dose Response in Commitant Esotropic Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham Yahya Abdel Mohsen AbdelHafez, Resident doctor, Assiut University
Other Study IDs: Medial rectus tendon width
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Strabismus
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Caliper — Measure medial rectus tendon width with caliper intraoperative

SUMMARY:
This study aims to investigate the clinical correlation between medial rectus tendon width and surgical dose response in esotropic patients undergoing medical rectus recession

DETAILED DESCRIPTION:
Esotropia is a type of strabismus where one or both eyes turn inward(1).Medial rectus tendon width is horizontal thickness of the tendon of the medial rectus muscle, one of the extraocular muscles.Medial rectus recession is a standard surgical treatment for esotropia involving weakening the medial rectus muscle by repositioning it posteriorly(2).Surgical Dose Response describes how much eye alignment in prism diopters is achieved per millimeter of muscle recession.

Studies on medial rectus resection revealed that higher medial rectus tendon width (MRTW) was associated with a larger surgical dose-response(3).Other studies revealed that the effect of lateral rectus recession in patients with intermittent exotropia was larger in cases with narrower lateral rectus tendon width (4,5).

The potential impact of medial rectus tendon width on the effectiveness of medial rectus recession had not been studied.

ELIGIBILITY:
Inclusion Criteria:

- All patients with comitant esotropia scheduled for unilateral or bilateral medial rectus recession

Exclusion Criteria:

* previous extraocular muscle surgery Incomitant esotropia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with comitant esotropia scheduled for unilateral or bilateral medial rectus recession
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Clinical correlation between medial rectus tendon width and surgical dose response in comitant esotropic patients undergoing medial rectus recession | Baseline
  Can medial rectus tendon width affect surgical dose response in commitant esotropic patients undergoing medial rectus recession
Variation in medial rectus tendon width in different age groups | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ali Natag Riad, Professor, Study Director — Assiut University; Mohammed Anwr Sayed, Assistant professor, Study Director — Assiut University; Sara Hussein AlAttar, Assistant professor, Study Director — Assiut University

REFERENCES:
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC3194326/
- See also: Related Info — https://www.nature.com/articles/6702002.pdf
- See also: Related Info — https://www.nature.com/articles/eye2009113